CLINICAL TRIAL: NCT06175494
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Clinical Study to Evaluate the Efficacy, Safety, and Immunogenicity of Booster Vaccination With Recombinant COVID-19 (XBB) Trimer Protein Vaccine (Sf9 Cell) for the Prevention of SARS-CoV-2 Infection in a Population of 18 Years of Age and Older.
Brief Title: A Phase 3 Clinical Study to Evaluate the Efficacy, Safety and Immunogenicity of Booster Vaccination With Recombinant COVID-19 (XBB) Trimer Protein Vaccine (Sf9 Cell)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Collaborators: WestVac Biopharma (Guangzhou) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WSKCT018
Record Dates: First submitted 2023-12-18; First posted 2023-12-19 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Recombinant COVID-19 (XBB) Trimer Protein Vaccine (Sf9 Cell)
  Interventions: Biological: Recombinant COVID-19 (XBB) Trimer Protein Vaccine (Sf9 Cell)
- Control group (Active Comparator): Recombinant COVID-19 Variant Vaccine（ Sf9 Cell）
  Interventions: Biological: Recombinant COVID-19 Variant Vaccine (Sf9 Cell)
- Placebo control group (Placebo Comparator): Placebo control
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant COVID-19 (XBB) Trimer Protein Vaccine (Sf9 Cell) — boost with Recombinant COVID-19 (XBB) Trimer Protein Vaccine (Sf9 Cell)
  Arms: Experimental group
Biological: Recombinant COVID-19 Variant Vaccine (Sf9 Cell) — boost with Recombinant COVID-19 Variant Vaccine (Sf9 Cell)
  Arms: Control group
Biological: Placebo — boost with saline
  Arms: Placebo control group

SUMMARY:
The Recombinant COVID-19 (XBB) Trimer Protein Vaccine (Sf9 Cell) developed by WestVac Biopharma Co., Ltd. is a monovalent modified vaccine designed against Omicron XBB.1.5.

This is a multi-center, randomized, double-blind, placebo-controlled phase 3 clinical study with two cohorts, i.e. the immuno-bridging observational cohort and the efficacy observational cohort, aims to evaluate the efficacy, safety, and immunogenicity of booster vaccination with Recombinant COVID-19 (XBB) Trimer Protein Vaccine (Sf9 Cell) for the prevention of SARS-CoV-2 infection in a population of 18 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years and above, including those with underlying diseases or immunocompromised.
2. Basic or booster vaccination with COVID-19 vaccine ≥3 months.
3. No history of SARS-CoV-2 infection history within 3 months, or never infected.
4. Have the ability to understand research procedures, with informed consent, voluntarily sign informed consent form, and be able to comply with the requirements of clinical study protocol.

Exclusion Criteria:

1. Axillary temperature ≥37.3℃.
2. SARS-CoV-2 antigen or nucleic acid screening positive during the screening period.
3. Anti-SARS-CoV-2 IgM antibody screening positive during the screening period.
4. It is in the advanced stage of malignant tumor and the disease control is unstable.
5. Female pregnancy (pregnancy test results are positive), lactation period.
6. Suffering from serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, heart failure etc.; suffering from severe hypertension that can not be controlled by drugs.
7. Suffering from other serious chronic conditions such as uncontrolled asthma, diabetes, chronic obstructive pulmonary disease, pulmonary embolism, chronic kidney disease requiring dialysis, cirrhosis of the liver, convulsions, epilepsy and other neurological/psychiatric conditions.
8. Have been diagnosed with congenital or acquired immunodeficiency, HIV infection (including anti-HIV antibody positive during the screening period).
9. People who are allergic to any component of the investigational vaccine and have a history of severe allergies or vaccine allergic reactions in the past.
10. Congenital or acquired angioedema/neuropathic edema.
11. Asplenia or functional asplenia.
12. Thrombocytopenia or other clotting disorders (which may cause intramuscular injection contraindications).
13. Received another investigational drug within 1 month prior to receiving the investigational vaccine.
14. Received subunit or inactivated vaccine within 14 days prior to receiving the investigational vaccine, or received live attenuated vaccine within 1 month.
15. Fertile female subjects did not use effective contraception within 1 month prior to enrollment.
16. Fertile female and male subjects have pregnancy plans and sperm/egg donation plans from the screening period to 3 months after vaccination.
17. Medical, psychological, social, or other conditions that, in the investigator's judgment, are inconsistent with the protocol or affect the subject's signing of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy against COVID-19 | 14 days to 6 months after vaccination
  Efficacy against the first occurrence of etiologically confirmed (antigen or PCR-positive) cases of symptomatic COVID-19, regardless of severity, 14 days to 6 months after booster vaccination.
AEs and ARs | 0-7 days after vaccination
  Incidence of adverse events (AEs) and adverse reactions (ARs) 0-7 days after booster vaccination.

SECONDARY OUTCOMES:
Efficacy against COVID-19 | 14 days to 6 months after booster vaccination
  Efficacy against the first occurrence of etiologically confirmed (antigen or PCR-positive) cases of moderate/severe COVID-19 caused by SARS-CoV-2 infection, cases of hospitalization due to COVID-19, and cases of death due to COVID-19, > 14 days to 6 months after booster vaccination.
Efficacy against COVID-19 | 7 days to 6 months after booster vaccination
  Efficacy against the first occurrence of etiologically confirmed (antigen or PCR-positive) cases of symptomatic COVID-19, regardless of severity, 7 days to 6 months after booster vaccination.
Efficacy against COVID-19 | 7 days to 6 months after booster vaccination
  Efficacy against the first occurrence of etiologically confirmed (antigen or PCR-positive) cases of moderate/severe COVID-19 caused by SARS-CoV-2 infection, cases of hospitalization due to COVID-19, and cases of death due to COVID-19, > 7 days to 6 months after booster vaccination.
AEs and ARs | 0-30 days after booster vaccination
  Incidence of adverse events (AEs) and adverse reactions (ARs) 0-30 days after booster vaccination.
SAEs and AESIs | within 12 months after booster vaccination
  Incidence of serious adverse events (SAE) and adverse events of special interest (AESI) within 12 months after booster vaccination.
Immunogenicity | day 14 after booster vaccination
  The geometric mean titer (GMT), seroconversion rate and geometric mean fold increase (GMI) of neutralizing antibodies (true virus and pseudo-virus assay) against SARS-CoV-2 Omicron XBB.1.5 variant and the main circulating strain at that time on day 14 after booster vaccination.
Immunogenicity | day 14, day 30, 3 months and 6 months after booster vaccination
  The geometric mean titer (GMT), seroconversion rate and geometric mean fold increase (GMI) of neutralizing antibodies (pseudo-virus assay) against SARS-CoV-2 Omicron XBB.1.5 variant and the main circulating strain at that time on day 14, day 30, 3 months and 6 months after booster vaccination.
Immunogenicity | day 14, day 30, 3 months and 6 months after booster vaccination
  The geometric mean titer (GMT), seroconversion rate and geometric mean fold increase (GMI) of IgG antibodies against SARS-CoV-2 S-RBD protein on day 14, day 30, 3 months and 6 months after booster vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Medical, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China